CLINICAL TRIAL: NCT06780579
Title: Expanded Access Treatment Protocol for Bulevirtide
Brief Title: Expanded Access for Bulevirtide
Status: Available | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-589-7094
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis Delta Virus Infection
MeSH Terms: interventions — bulevirtide

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Bulevirtide — 10 mg BLV will be administered via subcutaneous injection
  Other Names: GS-4438; Hepcludex®

SUMMARY:
The goal of this study is to provide access to bulevirtide (BLV (GS-4438), Hepcludex®) to eligible participants with chronic hepatitis delta virus infection (CHD).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with CHD as confirmed by medical records.
* Compensated liver disease with liver cirrhosis (defined by biopsy, Fibroscan, or clinically by the treating physician) and Child-Pugh score ≤ 6.
* Positive HDV RNA test within 6 months of initial EAP request (only applicable to patients who have not received treatment with BLV).

Key Exclusion Criteria:

* Coinfection with hepatitis C virus (HCV) (HCV viremia defined by polymerase chain reaction (PCR)) or uncontrolled HIV infection (CD4 < 500 cells/mm^3 and detectable HIV RNA).
* Current or previous (within last 3 months from screening) decompensated liver disease, including coagulopathy, hepatic encephalopathy, and esophageal varices hemorrhage.
* Significant medical diseases or conditions, that might decrease the benefit-risk ratio of participating in this program to an unacceptable level, as determined by the treating physician.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences

REFERENCES:
- [Derived] Mageras A, Rodriguez N, Katzenstein C, Lee F, Alpert L, Branch AD, Zhang X, Dieterich DT, Kushner T. Novel Implementation of Hepatitis B to Hepatitis Delta Reflex Testing in a US Healthcare System. Am J Gastroenterol. 2025 Jul 31. doi: 10.14309/ajg.0000000000003688. Online ahead of print. PMID 40736690